CLINICAL TRIAL: NCT04746300
Title: imPlementing ROutine Molecular Characterization in Patients With Metastatic Castration-resistant ProsTate Cancer by Next Generation DNA Sequencing (PROMPT-study)
Brief Title: imPlementing ROutine Molecular Characterization in Patients With Metastatic Castration Resistant ProstaTe Cancer by NGS
Acronym: PROMPT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: VGZ health insurance (NL) (Unknown); Paul Speth Foundation (NL) (Unknown); Radboud Oncology Fund (NL) (Unknown)
Responsible Party: Sponsor
Other Study IDs: MOURO41 - PROMPT; NL68315.091.19 (Registry Identifier: ABR registry)
Record Dates: First submitted 2021-01-28; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Prostate Cancer
Keywords: mCRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — CT-guided biopsies from lymph node, soft tissue, viscera and bone are collected. Blood and urine specimens are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: no sequencing: Participants in this group, for which DNA sequencing could not be reported due to a variety of (quality/technical) reasons, will be treated with standard of care therapy. This group is therefore comparable to patients treated outside the Radboudumc.
  Interventions: Procedure: Biopsy; Procedure: Blood sample
- Group 2: no druggable aberration: Participants in this group received a DNA sequencing report identifying no biomarkers to which a logical treatment option can be connected. These participants will also receive standard of care therapy.
  Interventions: Procedure: Biopsy; Procedure: Blood sample
- Group 3: allocated to personalized treatment: Participants in this group received a DNA sequencing report which identified presence of a biomarker allowing the participant to be treated with a personalized therapy. This therapy could range from immunotherapy, or PARP inhibitors, to other medication.
  Interventions: Procedure: Biopsy; Procedure: Blood sample

INTERVENTIONS:
Procedure: Biopsy — A biopsy will be taken from metastatic tissue, which will be used for DNA sequencing
Procedure: Blood sample — Blood samples will be taken for additional translational research

SUMMARY:
The PROMPT study aims to routinely implement genomic pre-sorting of metastatic castration-resistant prostate cancer (mCRPC) patients for personalized treatment (e.g. immuno-, PARP inhibitors, or platinum-therapy). The investigators hypothesize that, by doing this early in the disease course (before exhausting standard of care options), it will improve treatment planning, patient outcome, quality of life, and reduce costs.

DETAILED DESCRIPTION:
Prostate cancer is a major health problem leading to significant morbidity and mortality in men worldwide. Approved therapies for metastatic castration-resistant prostate cancer (mCRPC) include abiraterone and enzalutamide (targeting the androgen signaling pathway), radium-223 (bone targeting radionuclide therapy), and taxane chemotherapy. Controversy remains on optimal sequencing of available therapeutic agents, and these drugs are still commonly prescribed in a trial-and-error manner. Only a minority of patients receives the full benefit of the anticancer armamentarium, but all experience unnecessary side-effects, quality of life deterioration, and delay in onset to adequate life-prolonging treatment. In addition, the prescription of ineffective drugs and avoidable hospital admissions contribute to the financial burden of health care systems.

In recent years, distinct molecular subsets of prostate cancer have been identified in mCRPC. These molecular defects may guide physicians in proper sequencing of medication and in predicting the individual response more accurately. In previous studies using next-generation sequencing (NGS) mCRPC patients could be grouped into clearly distinct molecular subtypes. Moreover, in these subtypes biomarkers associated with resistance to certain therapies, or biomarkers actually predictive for enhanced response were identified.

In this study the investigators will introduce routine molecular characterization in participants with mCRPC as early as possible in their disease state. Participants will be screened before initiation of second-line treatment, since early identification will maximize clinical and financial benefit. Following screening, participants will be discussed in molecular tumor board and clinical meetings, and stratified to the agent they are most likely to respond to. Translational research is included to identify and validate additional predictive molecular biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 18 or older with adenocarcinoma of the prostate defined by: Documented histopathology at diagnosis of prostate adenocarcinoma without evidence of predominant or primary neuroendocrine histology.
2. Patients with a metastatic tumor site accessible for image-guided biopsy and allowing research analyses for this trial (e.g. biomarker testing by genomic, proteomic or transcriptomic assessment). A waiver can be made for patients presenting with metastatic hormone-sensitive prostate cancer (mHSPC), and no easily accessible tumour for biopsy and suitable primary tissue available for NGS.
3. Castration-resistant state (defined as disease progressing despite [chemical] castration per PCWG3 criteria)
4. Progressive disease as either

   * A rising PSA on minimum 2 serial consecutive measurements
   * Radiographic soft tissue progression per RECIST1.1 or bone progression per PCWG3 criteria
   * Clinical progression
5. At least one metastatic lesion present at baseline CT, MRI, 68Ga/18F-PSMA PET or bone scan
6. ECOG Performance status 0 to 2
7. Serum testosterone on castration level
8. Adequate renal function:

   • MDRD-GFR ≥ 30 ml/min/1.73m2
9. Adequate bone marrow function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x109/L
   * Hemoglobin (Hb) ≥ 5.6 mmol/L
10. Adequate liver function:

    * Total bilirubin level ≤ 2 institutional upper limit of the normal (ULN)
    * Aspartate aminotransferase (ASAT) ≤ 3 x ULN (or ≤ 5x ULN in case of known liver metastases)
    * Alanine aminotransferase (ALAT) ≤ 3 x ULN (or ≤ 5x ULN in case of known liver metastases)
11. Estimated life expectancy > 12 months
12. Willing and able to comply to the research protocol
13. Signed, written informed consent

Exclusion Criteria:

1. Prior chemotherapy and androgen receptor inhibition therapy related to castration resistant prostate cancer (one line of chemotherapy or androgen receptor inhibition may be given in the hormone-sensitive setting)
2. Active malignancy other than prostate cancer, except for patients with basal or squamous skin cancer. A waiver may be obtained from the PI in cases where the active malignancy is indolent and believed not to reduce mortality.
3. Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI).
4. Concurrent illness, including severe infection that may jeopardize the ability of the participant to undergo the procedures outlined in this protocol with reasonable safety
5. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse
6. Any condition which, in the opinion of the investigator, would preclude participation in this observational study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 600 patients with metastatic castration-resistant prostate cancer with clinical, radiographic or biochemical disease progression may be included in this study. The expected number of patients eligible for the protocol is well above 200 patients per year, including referrals from regional/community hospitals.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Responsiveness ratio | Throughout completion of study (estimated 5 years from start)
  Ratio of radiographic progression-free survival of personalized treatment or standard of care to the standard last line therapy (PFS-MPT-ratio vs PFS-SOC-ratio)

SECONDARY OUTCOMES:
Efficacy endpoint: ORR | Throughout completion of study (estimated 5 years from start)
  Best objective response rate (ORR) per RECIST1.1 criteria
Efficacy endpoint: rPFS | Throughout completion of study (estimated 5 years from start)
  Radiographic progresssion free survival (per RECIST1.1)
Efficacy endpoint: PSA response | Throughout completion of study (estimated 5 years from start)
  PSA decline >50% at 12 weeks or later
Efficacy endpoint: PSA-PFS | Throughout completion of study (estimated 5 years from start)
  Time to PSA progression (per PCWG3 criteria)
Efficacy endpoint: OS | Throughout completion of study (estimated 5 years from start)
  Overall survival capped at 1 year
Quality of life endpoint: EORTC-QLQ-30 | Throughout completion of study (estimated 5 years from start)
  Score of EORTC-QLQ-30 questionnaire
Quality of life endpoint: EPIC-26 | Throughout completion of study (estimated 5 years from start)
  Score of EPIC-26 questionnaire
Quality of life endpoint: EQ-5D-5L | Throughout completion of study (estimated 5 years from start)
  Score of EQ-5D-5L questionnaire
Quality of life endpoint: BIP-SF | Throughout completion of study (estimated 5 years from start)
  Score of BIP-SF questionnaire
Medical Resource Utilization (MRU); nr of lines | At the end of year 1, year 2, year 3, and at completion of the study (estimated end of year 5)
  Averaged number of lines of standard care per year
Medical Resource Utilization (MRU); costs | At the end of year 1, year 2, year 3, and at completion of the study (estimated end of year 5)
  Averaged costs of standard care per year
Medical Resource Utilization (MRU); treatment-related costs | At the end of year 1, year 2, year 3, and at completion of the study (estimated end of year 5)
  Averaged costs of treatment-related resource utilization (e.g. admissions in ward or ICU) per admission and/or per duration

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud UMC, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided